CLINICAL TRIAL: NCT00910026
Title: Exhaled Breath Condensate (EBC) Collection and Analysis in Mechanically Ventilated ICU Patients: Monitoring of the Influence of Various Tidal Volumes on Lung Inflammatory Biomarkers
Brief Title: Study of the Influence of Various Tidal Volumes on Exhaled Breath Condensate (EBC) in Mechanically Ventilated Patients
Acronym: TDEBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Apostolopoulou Olympia, MD, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4163/02-09-2008
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2009-11

CONDITIONS: Inflammation
Keywords: EBC and mechanical ventilation; low tidal volume ventilation; high tidal volume ventilation; inflammatory and oxidative stress EBC biomarkers; Ventilator induced lung injury
MeSH Terms: conditions — Inflammation; Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- low tidal volume ventilation (Experimental): 6 ml/kg tidal volume ventilation
  Interventions: Procedure: low tidal volume ventilation
- high tidal volume ventilation (Experimental): 12 ml/kg tidal volume ventilation
  Interventions: Procedure: high tidal volume ventilation

INTERVENTIONS:
Procedure: low tidal volume ventilation — 6 ml/kg tidal volume ventilation
  Arms: low tidal volume ventilation
Procedure: high tidal volume ventilation — 12 ml/kg tidal volume ventilation
  Arms: high tidal volume ventilation

SUMMARY:
The aim of the present study is to evaluate the effect of low (6 ml/kg) and high (12 ml/kg) tidal volume ventilation on inflammatory and oxidative stress biomarkers in the exhaled breath condensate (EBC) of ICU patients without lung injury. As the analysis of EBC is reflecting the composition of epithelial lining fluid (ELF), the study of EBC pH and inflammatory and oxidative stress markers could have the potential for assessing lung inflammation caused by mechanical ventilation. This study also aims to look at the possibility to identify selective profiles of biomarkers that might have a prognostic and/or diagnostic value in the follow up of these patients.

DETAILED DESCRIPTION:
INTRODUCTION:

Airway inflammation plays a key role in many airway diseases. Non invasive methods to study these inflammatory processes and to monitor airway diseases are in high demand. Stimulating interest is in breath analysis, such as the analysis of exhaled breath condensate (EBC), a technique of sampling the epithelial lining fluid of the lung (ELF), as an even easier way to assess airway inflammation (1,2). The appeal of EBC lies in its ability to collect non-invasively a wide range of nonvolatile molecules from the respiratory tract, the fact that it can be repeated frequently within short intervals without adverse events and that collection devices can be used in a wide range of settings including intensive care units (3,4,5,6).

Analysis of EBC could not be limited to patient monitoring and understanding mechanisms of pulmonary disease. It also could become a useful tool for monitoring and screening for healthy individuals for possible early pulmonary tissue damage (6,7). There is a special need for more data on intra-subject and day-to-day variation, both essential for the decision as to whether a biomarker can serve as a research tool or even has the potential for disease monitoring in clinical practice (7).

It has been recognized for some time that mechanical ventilation may induce lung injury and inflammation (8,9,10). Recent experimental and clinical data suggest that in healthy lungs, mechanical ventilation with tidal volume ranging between 7 and 12 ml/kg in the absence of positive end-expiratory pressure may lead to endothelial, extracellular matrix and peripheral airways damage without major inflammatory response, which further worsen with higher tidal volumes (15,34). Several mechanisms may explain damage to the lung structure induced by mechanical ventilation: regional over distension, 'low lung volume' associated with tidal airway closure, and inactivation of surfactant (15).

High tidal volume ventilation has been shown to result in increased mortality while low tidal volume ventilation is regarded as a lung protective strategy in ALI, ARDS (11,12,13,35).

In contrast, in other randomized studies (31,32) including a heterogeneous group of major thoracic and abdominal surgical procedures, protective mechanical ventilation was not associated with a decrease in intrapulmonary and systemic inflammation. Furthermore, there was no evidence that protective ventilation prevented lung adverse effect or decreased systemic cytokine levels in cardiac surgery (33).

In line with these observations and considering that a practical parameter of increased mechanical stress of the lung remains to be demonstrated, studies may address the question whether the analysis of EBC biomarkers are related to ventilator-induced lung injury by low or high tidal volumes.

MATERIALS AND METHODS:

The present study is a prospective, randomized, controlled trial that will take place in the ICU of the University Hospital of Larissa, Thessaly. Authorization has been given from the Scientific Council and the ethical committee of our hospital.

Patients:

ICU patients requiring mechanical ventilation because of stroke, subarachnoid and/or intracerebral hemorrhage and with healthy respiratory system (evaluated using criteria as the LISS - Murray Lung Injury Severity Score) (14).

Interventions:

EBC collection will be performed on mechanically ventilated patients through the endotracheal tube according to ATS/ERS task force 2005 (7). Patients must be hemodynamically and respiratory stable.

All patients will be under sedation and will receive ventilation by volume control. The respiratory frequency will be adapted at the set tidal volume in order to maintain the pH values within normal limits (7.35-7.45). SaO2 will be maintained equal or superior to 95%.

EBC will be collected by inserting a special conduit (FILT, lung and chest diagnostics Ltd. Berlin Germany) for the breath condensate collecting device (Ecoscreen, Jaeger, Germany) into the expiratory limb of the ventilator tubing. Collecting time for EBC will be 30 min. No humidification will be used during the collection.

The acidity (pH) of EBC before and after de-aeration with an inert gas Argon, 350 ml/minutes for 10 minutes, (gas standardisation) (17) will be readily measured using a pH meter Jenway Model 3510.

All samples will be stored at -80 ο C for subsequent mediator measurements. Variables of ventilation (frequency, PEEP, FIO2, Vt), lung mechanics, arterial pressure, heart rate, arterial blood saturation, ICP and gas blood samples examination will be registered before and during the EBC collection. Also will be registered indices of lung injury (PiO2/FiO2, LISS), indices of systemic inflammation (temperature, leucocyte and neutrophil counts in blood samples) during the observation period. Disease severity indices (SOFA, SAPS, APACHE II) will be registered during the initial assessment.

EBC analysis:

EBC collected will be analyzed for pH, 8-isoprostane, H2O2, nitrites/nitrates and cytokines. The measurement of biomarkers will be performed using standardized procedures, as previously described.

pH measurements: pH will be measured as previously described (16,17). H2O2 measurements: H2O2 concentration will be determined by an enzymatic assay using horseradish peroxidase (Sigma Chemicals, St. Louis, MO), as previously described (17,18,19,20).

8-Isoprostane measurements: 8-Isoprostane will be determined by a competitive enzyme immunoassay kit (Cayman Chemical, Ann Arbor, MI), as previously described (17,18,21,29). The detection limit of the assay is 4 pg/ml.

Nitrogen oxides, nitrite/nitrate (NO2/NO3), and related products measurements: will be performed as previously described (17,22). Briefly, will be determined by using spectrophotometric assays (Griess reaction) (23,24,25,26,27,28).

Cytokines measurement: will be quantified by EIA/ELISA kits as previously described (24,25,29,30).

Protocol Details:

The patients after the initial assessment will be randomized to receive mechanical ventilation with 6 or 12 ml/Kg of ideal body weight calculated through the following equation:

For men [(Height (cm)-154) x 0.9] +50 and For women [(Height (cm)-154) x 0.9] +45.5. The observation period will be a minimum of 10 days (if possible) and EBC collection will be performed within the first 24 hours of admission (day 0) and through the days 1,2,4,6,8,10.

EBC collection at day 0 will be performed under both modalities of ventilation with the purpose to investigate the quantity and composition of the collected EBC from the same patient ventilated with different tidal volumes. For the next measurements, the EBC collection for each group will be performed under the preset conditions of ventilation.

Complications such as VAP, ARDS or sepsis during the period of observation will be recorded.

Statistical analysis:

Analysis will be performed using SPSS for Windows v. 16.0. Normality of distribution will be checked with Kolmogorov-Smirnov test. Normally distributed data will be presented as mean ± standard deviation (SD), whereas skewed data as median (interquartile range). Comparisons between two groups will be evaluated with unpaired t tests for normally distributed and Mann-Whitney tests for skewed data. Comparisons between more than two groups will be performed with analysis of variance (ANOVA) with appropriate post hoc tests

ELIGIBILITY:
Inclusion Criteria:

* ICU patients mechanically ventilated because of stroke, subarachnoid and/or intracerebral hemorrhage
* Healthy respiratory system

Exclusion Criteria:

* Pulmonary diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of low (6 ml/kg) and high (12 ml/kg) tidal volume ventilation on inflammatory and oxidative stress biomarkers in the exhaled breath condensate (EBC) of ICU patients without lung injury. | 2 years

SECONDARY OUTCOMES:
Evaluation of the prognostic role of exhaled biomarkers in the subsequent outcome of mechanically ventilated patients (length of ICU hospitalization, subsequent development of ALI or ARDS and morbidity and mortality in the ICU). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olympia I. Apostolopoulou, MD, Principal Investigator — University of Thessaly
Locations (1):
- Intensive Care Unit Department of University Hospital of Larissa, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Holz O. Catching breath: monitoring airway inflammation using exhaled breath condensate. Eur Respir J. 2005 Sep;26(3):371-2. doi: 10.1183/09031936.05.00071305. No abstract available. PMID 16135713
- [Background] Hunt J. Exhaled breath condensate: an evolving tool for noninvasive evaluation of lung disease. J Allergy Clin Immunol. 2002 Jul;110(1):28-34. doi: 10.1067/mai.2002.124966. PMID 12110814
- [Background] Mutlu GM, Garey KW, Robbins RA, Danziger LH, Rubinstein I. Collection and analysis of exhaled breath condensate in humans. Am J Respir Crit Care Med. 2001 Sep 1;164(5):731-7. doi: 10.1164/ajrccm.164.5.2101032. No abstract available. PMID 11549524
- [Background] Kharitonov SA, Barnes PJ. Exhaled markers of pulmonary disease. Am J Respir Crit Care Med. 2001 Jun;163(7):1693-722. doi: 10.1164/ajrccm.163.7.2009041. No abstract available. PMID 11401895
- [Background] Muller WG, Morini F, Eaton S, Peters M, Jaffe A. Safety and feasibility of exhaled breath condensate collection in ventilated infants and children. Eur Respir J. 2006 Sep;28(3):479-85. doi: 10.1183/09031936.06.00063505. Epub 2006 Apr 26. PMID 16641124
- [Background] Moloney ED, Mumby SE, Gajdocsi R, Cranshaw JH, Kharitonov SA, Quinlan GJ, Griffiths MJ. Exhaled breath condensate detects markers of pulmonary inflammation after cardiothoracic surgery. Am J Respir Crit Care Med. 2004 Jan 1;169(1):64-9. doi: 10.1164/rccm.200307-1005OC. Epub 2003 Oct 9. PMID 14551168
- [Background] Horvath I, Hunt J, Barnes PJ, Alving K, Antczak A, Baraldi E, Becher G, van Beurden WJ, Corradi M, Dekhuijzen R, Dweik RA, Dwyer T, Effros R, Erzurum S, Gaston B, Gessner C, Greening A, Ho LP, Hohlfeld J, Jobsis Q, Laskowski D, Loukides S, Marlin D, Montuschi P, Olin AC, Redington AE, Reinhold P, van Rensen EL, Rubinstein I, Silkoff P, Toren K, Vass G, Vogelberg C, Wirtz H; ATS/ERS Task Force on Exhaled Breath Condensate. Exhaled breath condensate: methodological recommendations and unresolved questions. Eur Respir J. 2005 Sep;26(3):523-48. doi: 10.1183/09031936.05.00029705. PMID 16135737
- [Background] Thammanomai A, Majumdar A, Bartolak-Suki E, Suki B. Effects of reduced tidal volume ventilation on pulmonary function in mice before and after acute lung injury. J Appl Physiol (1985). 2007 Nov;103(5):1551-9. doi: 10.1152/japplphysiol.00006.2007. Epub 2007 Aug 9. PMID 17690203
- [Background] Halter JM, Steinberg JM, Gatto LA, DiRocco JD, Pavone LA, Schiller HJ, Albert S, Lee HM, Carney D, Nieman GF. Effect of positive end-expiratory pressure and tidal volume on lung injury induced by alveolar instability. Crit Care. 2007;11(1):R20. doi: 10.1186/cc5695. PMID 17302983
- [Background] Del Sorbo L, Slutsky AS. Year in review 2007: Critical Care--respirology. Crit Care. 2008;12(5):231. doi: 10.1186/cc6953. Epub 2008 Oct 14. PMID 18983706
- [Background] Dreyfuss D, Saumon G. From ventilator-induced lung injury to multiple organ dysfunction? Intensive Care Med. 1998 Feb;24(2):102-4. doi: 10.1007/s001340050529. No abstract available. PMID 9539065
- [Background] Parker JC, Hernandez LA, Peevy KJ. Mechanisms of ventilator-induced lung injury. Crit Care Med. 1993 Jan;21(1):131-43. doi: 10.1097/00003246-199301000-00024. PMID 8420720
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Murray JF, Matthay MA, Luce JM, Flick MR. An expanded definition of the adult respiratory distress syndrome. Am Rev Respir Dis. 1988 Sep;138(3):720-3. doi: 10.1164/ajrccm/138.3.720. No abstract available. PMID 3202424
- [Background] Pelosi P, Negrini D. Extracellular matrix and mechanical ventilation in healthy lungs: back to baro/volotrauma? Curr Opin Crit Care. 2008 Feb;14(1):16-21. doi: 10.1097/MCC.0b013e3282f25162. PMID 18195621
- [Background] Vaughan J, Ngamtrakulpanit L, Pajewski TN, Turner R, Nguyen TA, Smith A, Urban P, Hom S, Gaston B, Hunt J. Exhaled breath condensate pH is a robust and reproducible assay of airway acidity. Eur Respir J. 2003 Dec;22(6):889-94. doi: 10.1183/09031936.03.00038803. PMID 14680074
- [Background] Kostikas K, Papatheodorou G, Ganas K, Psathakis K, Panagou P, Loukides S. pH in expired breath condensate of patients with inflammatory airway diseases. Am J Respir Crit Care Med. 2002 May 15;165(10):1364-70. doi: 10.1164/rccm.200111-068OC. PMID 12016097
- [Background] Kostikas K, Papatheodorou G, Psathakis K, Panagou P, Loukides S. Oxidative stress in expired breath condensate of patients with COPD. Chest. 2003 Oct;124(4):1373-80. doi: 10.1378/chest.124.4.1373. PMID 14555568
- [Background] van Beurden WJ, Harff GA, Dekhuijzen PN, van den Bosch MJ, Creemers JP, Smeenk FW. An efficient and reproducible method for measuring hydrogen peroxide in exhaled breath condensate. Respir Med. 2002 Mar;96(3):197-203. doi: 10.1053/rmed.2001.1240. PMID 11908513
- [Background] Razola SS, Ruiz BL, Diez NM, Mark HB Jr, Kauffmann JM. Hydrogen peroxide sensitive amperometric biosensor based on horseradish peroxidase entrapped in a polypyrrole electrode. Biosens Bioelectron. 2002 Dec;17(11-12):921-8. doi: 10.1016/s0956-5663(02)00083-0. PMID 12392940
- [Background] Montuschi P, Collins JV, Ciabattoni G, Lazzeri N, Corradi M, Kharitonov SA, Barnes PJ. Exhaled 8-isoprostane as an in vivo biomarker of lung oxidative stress in patients with COPD and healthy smokers. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1175-7. doi: 10.1164/ajrccm.162.3.2001063. PMID 10988150
- [Background] Ganas K, Loukides S, Papatheodorou G, Panagou P, Kalogeropoulos N. Total nitrite/nitrate in expired breath condensate of patients with asthma. Respir Med. 2001 Aug;95(8):649-54. doi: 10.1053/rmed.2001.1117. PMID 11530952
- [Background] 23. Hammerschmidt S., Meybaum M., Schauer J. et. al; Effect of tidal volume and end expiratory pressure on pulmonary NO release in an isolated lung model (abstract); Eur.Respir.J. 2001;18(suppl):366s.
- [Background] Berg JT, Deem S, Kerr ME, Swenson ER. Hemoglobin and red blood cells alter the response of expired nitric oxide to mechanical forces. Am J Physiol Heart Circ Physiol. 2000 Dec;279(6):H2947-53. doi: 10.1152/ajpheart.2000.279.6.H2947. PMID 11087251
- [Background] Francoeur C, Denis M. Nitric oxide and interleukin-8 as inflammatory components of cystic fibrosis. Inflammation. 1995 Oct;19(5):587-98. doi: 10.1007/BF01539138. PMID 8543373
- [Background] Jang AS, Choi IS, Lee S, Seo JP, Yang SW, Park KO, Lee KY, Lee JU, Park CS, Park HS. Nitric oxide metabolites in induced sputum: a marker of airway inflammation in asthmatic subjects. Clin Exp Allergy. 1999 Aug;29(8):1136-42. doi: 10.1046/j.1365-2222.1999.00595.x. PMID 10457119
- [Background] Edwards YS, Sutherland LM, Murray AW. NO protects alveolar type II cells from stretch-induced apoptosis. A novel role for macrophages in the lung. Am J Physiol Lung Cell Mol Physiol. 2000 Dec;279(6):L1236-42. doi: 10.1152/ajplung.2000.279.6.L1236. PMID 11076814
- [Background] Gessner C, Hammerschmidt S, Kuhn H, Lange T, Engelmann L, Schauer J, Wirtz H. Exhaled breath condensate nitrite and its relation to tidal volume in acute lung injury. Chest. 2003 Sep;124(3):1046-52. doi: 10.1378/chest.124.3.1046. PMID 12970036
- [Background] Carpagnano GE, Kharitonov SA, Resta O, Foschino-Barbaro MP, Gramiccioni E, Barnes PJ. Increased 8-isoprostane and interleukin-6 in breath condensate of obstructive sleep apnea patients. Chest. 2002 Oct;122(4):1162-7. doi: 10.1378/chest.122.4.1162. PMID 12377837
- [Background] Sack U, Scheibe R, Wotzel M, Hammerschmidt S, Kuhn H, Emmrich F, Hoheisel G, Wirtz H, Gessner C. Multiplex analysis of cytokines in exhaled breath condensate. Cytometry A. 2006 Mar;69(3):169-72. doi: 10.1002/cyto.a.20231. PMID 16496377
- [Background] Wrigge H, Uhlig U, Zinserling J, Behrends-Callsen E, Ottersbach G, Fischer M, Uhlig S, Putensen C. The effects of different ventilatory settings on pulmonary and systemic inflammatory responses during major surgery. Anesth Analg. 2004 Mar;98(3):775-81, table of contents. doi: 10.1213/01.ane.0000100663.11852.bf. PMID 14980936
- [Background] Wrigge H, Zinserling J, Stuber F, von Spiegel T, Hering R, Wetegrove S, Hoeft A, Putensen C. Effects of mechanical ventilation on release of cytokines into systemic circulation in patients with normal pulmonary function. Anesthesiology. 2000 Dec;93(6):1413-7. doi: 10.1097/00000542-200012000-00012. PMID 11149435
- [Background] Koner O, Celebi S, Balci H, Cetin G, Karaoglu K, Cakar N. Effects of protective and conventional mechanical ventilation on pulmonary function and systemic cytokine release after cardiopulmonary bypass. Intensive Care Med. 2004 Apr;30(4):620-6. doi: 10.1007/s00134-003-2104-5. Epub 2004 Jan 13. PMID 14722635
- [Background] Bonetto C, Terragni P, Ranieri VM. Does high tidal volume generate ALI/ARDS in healthy lungs? Intensive Care Med. 2005 Jul;31(7):893-5. doi: 10.1007/s00134-005-2668-3. Epub 2005 Jun 2. No abstract available. PMID 15931524
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162